CLINICAL TRIAL: NCT02270268
Title: Therapeutic Effects of Pectin Supplementation in Patients With Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: Effects of Pectin Supplementation in Diarrhea-predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Nanjing PLA General Hospital, Nanjing PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011NLY073
Record Dates: First submitted 2014-10-10; First posted 2014-10-21 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Gut microbiota; Soluble dietary fiber
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Pectins; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pectin (Experimental): a kind of soluble dietary fiber
  Interventions: Dietary Supplement: Pectin
- Placebo (Placebo Comparator): maltodextrin
  Interventions: Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: Pectin — Pectin （Andeli Ltd. Yantai, China）, 24g/d for six weeks
  Arms: pectin
Dietary Supplement: maltodextrin
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of pectin, a kind of soluble dietary fiber, on clinical symptoms, gut microbiota and the immune status in patients with diarrhea-predominant irritable bowel syndrome

DETAILED DESCRIPTION:
Patients were randomized to receive either pectin or placebo. Treatment consisted of 6 weeks supplementation with pectin (fiber group) or placebo (maltodextrin). We evaluated the clinical symptoms, gut microbiota and the immune markers in two groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients(age≧18y)
* Admitted for diarrhea-predominant irritable bowel syndrome

Exclusion Criteria:

* Mental disorders
* Cancer
* Inflammatory bowel disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
efficacy: change of stool frequency, faecal form and clinical symptoms score | six weeks after inclusion
  change from baseline in stool frequency, faecal form (Bristol stool scale) and clinical symptoms score (7-point Likert scale) at six weeks

SECONDARY OUTCOMES:
efficacy: gut microbiota | six weeks after inclusion
  real-time PCR
efficacy: cytokine ratios | six weeks after inclusion
  Cytokine production

CONTACTS AND LOCATIONS:
Overall Officials: Tao Gao, M.D., Principal Investigator — Nanjing PLA General Hospital